CLINICAL TRIAL: NCT00088465
Title: An Open-Label Study of Intramuscular Olanzapine Depot in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Open-Label Study of Intramuscular Olanzapine Depot in Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5995; F1D-MC-HGKB (Other: Eli Lilly and Company)
Record Dates: First submitted 2004-07-26; First posted 2004-07-27 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Schizophrenic Disorders; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

ARMS (1):
- Intramuscular Olanzapine Depot (Experimental): Intramuscular (IM) olanzapine depot flexible dosing and flexible interval
  Interventions: Drug: Intramuscular olanzapine depot

INTERVENTIONS:
Drug: Intramuscular olanzapine depot — 45-405 milligram (mg), intramuscular injection, on a 2-, 3-, or 4-week interval.
  Other Names: LY170053; Zyprexa Adhera

SUMMARY:
This is a long-term, open-label clinical study designed to enable longer-term treatment of patients completing other clinical studies with intramuscular olanzapine depot.

Key objectives of the study are to:

* Determine how well intramuscular (IM) olanzapine depot works during long-term treatment,
* Evaluate the safety and tolerability of IM olanzapine depot during long-term treatment,
* Determine the blood levels of IM olanzapine depot in patients during long-term treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients must have schizophrenia
* Female patients of childbearing potential must be using a medically accepted means of contraception
* Patients must have completed (within 10 days) another IM olanzapine depot study if permitted by that study's protocol.

Exclusion Criteria:

* Patients must not have participated in a clinical trial of another investigational drug, including olanzapine, within 1 month (30 days) prior to study entry
* Female patients must not be pregnant or breast-feeding
* Patients must not be experiencing acute, serious or unstable medical conditions other than schizophrenia or schizoaffective disorder
* Patients must not have a substance (except nicotine or caffeine) dependence within the past 30 days

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 931 (Actual)
Dates: Start 2004-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (92):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Ana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bradenton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chagrin Falls, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chardon, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kirkland, Washington
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lanús Este
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mendoza
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glenside, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dandenong, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Diest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aparecida de Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb, Croatia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague, Czechia
- France (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayonne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bourg-en-Bresse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dole
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fontaine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Foron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Seyne-sur-Mer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Narbonne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Cyr-au-Mont-d'Or
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suresnes
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Saarow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest, Hungary
- Israel (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beer Yaacov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hod HaSharon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lev Hasharon
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savigliano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Enschede
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Hague
- Poland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
- Portugal (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Puerto Rico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mayagüez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava, Slovakia
- South Africa (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Randburg
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burgos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- [Derived] McDonnell DP, Landry J, Detke HC. Long-term safety and efficacy of olanzapine long-acting injection in patients with schizophrenia or schizoaffective disorder: a 6-year, multinational, single-arm, open-label study. Int Clin Psychopharmacol. 2014 Nov;29(6):322-31. doi: 10.1097/YIC.0000000000000038. PMID 24850228
- [Derived] Atkins S, Detke HC, McDonnell DP, Case MG, Wang S. A pooled analysis of injection site-related adverse events in patients with schizophrenia treated with olanzapine long-acting injection. BMC Psychiatry. 2014 Jan 14;14:7. doi: 10.1186/1471-244X-14-7. PMID 24423017
- [Derived] Peuskens J, Porsdal V, Pecenak J, Handest P, D'yachkova Y, Brousil R, Deberdt W. Schizophrenia symptoms and functioning in patients receiving long-term treatment with olanzapine long-acting injection formulation: a pooled analysis. BMC Psychiatry. 2012 Aug 31;12:130. doi: 10.1186/1471-244X-12-130. PMID 22935168
- [Derived] McDonnell DP, Detke HC, Bergstrom RF, Kothare P, Johnson J, Stickelmeyer M, Sanchez-Felix MV, Sorsaburu S, Mitchell MI. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, II: investigations of mechanism. BMC Psychiatry. 2010 Jun 10;10:45. doi: 10.1186/1471-244X-10-45. PMID 20537130
- [Derived] Detke HC, McDonnell DP, Brunner E, Zhao F, Sorsaburu S, Stefaniak VJ, Corya SA. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, I: analysis of cases. BMC Psychiatry. 2010 Jun 10;10:43. doi: 10.1186/1471-244X-10-43. PMID 20537128

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intramuscular Olanzapine Depot
Started | 931
Completed | 370
Not Completed | 561
Not completed — Withdrawal by Subject | 290
Not completed — Adverse Event | 77
Not completed — Lost to Follow-up | 57
Not completed — Physician Decision | 45
Not completed — Sponsor Decision | 37
Not completed — Lack of Efficacy | 27
Not completed — Protocol Violation | 17
Not completed — Death | 11

BASELINE CHARACTERISTICS:
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
Age Continuous [Mean (Standard Deviation); unit: years] | 39.32 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310
  Male | 621
Race/Ethnicity, Customized [Number; unit: participants]
  African | 102
  Caucasian | 629
  East Asian | 39
  Hispanic | 140
  Native American | 2
  West Asian | 19
Region of Enrollment [Number; unit: participants]
  United States | 177
  Portugal | 18
  Taiwan | 30
  Slovakia | 13
  Spain | 24
  Russian Federation | 114
  Israel | 29
  Italy | 6
  France | 55
  Puerto Rico | 27
  Australia | 11
  South Africa | 28
  Netherlands | 8
  Austria | 10
  Czech Republic | 3
  Hungary | 13
  Mexico | 63
  Argentina | 73
  Poland | 33
  Brazil | 89
  Belgium | 13
  Croatia | 16
  Romania | 34
  Germany | 32
  Sweden | 9
  Greece | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: The list of serious adverse events (SAE) and other non-serious adverse events (AE) are in Adverse Events Section.
Time Frame: Randomization to end of study up to 76 months
Population: All randomized participants who took at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
participants
  AE | 501
  SAE | 170

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Scores at Month 76 Endpoint
Description: Assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210.
Time Frame: Baseline, up to 76 months
Population: Participants with a baseline measurement and at least one post-baseline measurement, last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 856
units on a scale | 0.30 (16.42)

3. Secondary Outcome: Change From Baseline in PANSS Positive Scores at Month 76 Endpoint
Description: PANSS questions 1-7. Assesses positive symptoms associated with schizophrenia. 7 items make up the positive scale (ex. delusions, conceptual disorganization, and hallucinatory behavior). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total positive subscale scores range from 7 to 49.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 856
units on a scale | 0.21 (4.69)

4. Secondary Outcome: Change From Baseline in PANSS Negative Scores at Month 76 Endpoint
Description: PANSS questions 8-14. Assesses negative symptoms associated with schizophrenia. 7 items make up the negative scale (e.g. blunted affect, emotional withdrawal, poor rapport, and passive/apathetic social withdrawal). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total negative subscale scores range from 7 to 49.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 856
units on a scale | -0.08 (5.14)

5. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscales at Month 76 Endpoint
Description: PANSS General Psychopathology Subscale is the Remaining 16 PANSS questions or PANSS Question15 through Question 30. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 16 items is defined as the PANSS General Psychopathology Subscales. Possible score ranges from 16 to 112.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 856
units on a scale | 0.19 (8.51)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity of Illness (CGI-S) Scores at Month 72 Endpoint
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, up to 72 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 920
units on a scale | -0.17 (0.03)

7. Secondary Outcome: Change From Baseline in the Heinrichs-Carpenter Quality of Life Scale (QLS) Total Score at Month 76 Endpoint
Description: Heinrich-Carpenter QLS is an interviewer-rated scale which measures the impact of negative symptoms on occupational, social, and psychological functioning in patients with schizophrenia or schizoaffective disorder. Each of 21 items is rated on a scale from 0 (severely impaired functioning) to 6 (normal or adequate functioning), for a total score range of 0-126. Results are presented as change in Total score.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 852
units on a scale | 6.75 (18.55)

8. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) at Month 76 Endpoint
Description: A self-reported questionnaire that consists of 36 questions covering 8 health domains (physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. The mental component summary (MCS) and the physical component summary (PCS) have been constructed based on the 8 SF-36 domains.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 850
units on a scale
  Mental component summary | 0.94 (11.05)
  Physical component summary | -0.36 (8.34)

9. Secondary Outcome: Number of Psychiatric Visits
Description: Psychiatric visits were outpatient visits to a psychiatrist or psychiatric nurse.
Time Frame: Randomization to end of study up to 76 months
Population: All randomized participants who took at least one dose of study drug.
Measure: Number; unit: visits
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
visits | 14102

10. Secondary Outcome: Days of Hospitalization
Description: This is the total number of days for all hospitalized patients that were admitted to General, Psychiatric Ward as well as Intensive Care Unit (ICU).
Time Frame: Randomization to end of study up to 76 months
Population: All randomized participants who took at least one dose of study drug.
Measure: Number; unit: days
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
days
  Regular hospital | 2386
  Psychiatric hospital | 35587
  ICU | 134

11. Secondary Outcome: Change From Baseline in the Subjective Well-Being Under Neuroleptic Treatment-Short Form (SWN-S) at Month 76 Endpoint
Description: The Subjective Well-Being under Neuroleptic Treatment-Short Form (SWN-S) is a patient self-rated scale developed to measure the subjective well-being for the previous 7 days of a patient under neuroleptic treatment. The SWN-S consists of 20 items (each item is rated from 1=not at all to 6=very much). Possible total score ranges from 20-120.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 755
units on a scale | 0.86 (15.96)

12. Secondary Outcome: Patient Satisfaction With Medication Questionnaire-Modified (PSMQ) at Month 76 Endpoint
Description: Self-rated scale that measures patient's level of satisfaction with current antipsychotic medication. Consists of 3 items assessing satisfaction with current study medication (scored from 1='very dissatisfied' to 5='very satisfied'), preference comparing current study medication versus previous medications (scored from 1='much prefer previous medication' to 5='much prefer study medication'), and side effects of current study medication compared with previous medications (scored from 1='much less side effects' to 5='much more side effects'). Range of possible scores is 3-15.
Time Frame: Randomization to end of study up to 76 months
Population: All randomized participants.
Measure: Number; unit: percent of participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
percent of participants
  Depot, somewhat or very satisfied | 73.2
  Depot vs. oral, prefer or much prefer | 66.8
  Depot vs. oral, less or much less side effects | 73.3

13. Secondary Outcome: Plasma Olanzapine Concentrations in Participants During Long-Term Treatment by Year
Description: Plasma olanzapine concentrations are expressed as (nanogram/milliliter)/(milligram/day) ([ng/mL]/[mg/day]).
Time Frame: Randomization to end of study up to 76 months
Population: Participants who took at least one dose of study drug and had post-baseline measurements.
Measure: Mean (Standard Deviation); unit: (ng/mL)/(mg/day)
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
(ng/mL)/(mg/day)
  0.25 year (n= 130) | 2.23 (1.34)
  1 year (n= 189) | 2.51 (1.30)
  2 years (n= 166) | 2.45 (1.32)
  3 years (n= 148) | 2.65 (1.39)
  4 years (n= 109) | 2.57 (1.72)
  5 years (n= 87) | 2.59 (1.46)
  6 years (n= 28) | 2.73 (1.25)

14. Primary Outcome: Number of Participants With Treatment-Emergent Abnormal High Prolactin at Any Time Post Baseline
Description: Prolactin normal reference ranges for female: 2.0 - 29.0 nanograms per milliliter (ng/mL); male: 2.0 - 20.0 ng/mL. High value is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time after baseline.
Time Frame: Randomization to end of study up to 76 months
Population: Participants with normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 430
participants | 100

15. Primary Outcome: Number of Participants With Treatment-Emergent Abnormal High Alanine Transaminase (ALT), High Aspartate Transaminase (AST), High Total Bilirubin at Any Time Post Baseline
Description: High ALT is defined as a baseline value of <3 times the upper limit of normal (ULN) to ≥3 times the ULN at any time post baseline. High AST is defined as a baseline value of <5 times the ULN to ≥5 times the ULN at any time post baseline. High total bilirubin is defined as a baseline value of <2 times the ULN to ≥2 times the ULN at any time post baseline.
Time Frame: Randomization to end of study up to 76 months
Population: Participants with normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
participants
  ALT (n=901) | 61
  AST (n=909) | 55
  Total Bilirubin (n=912) | 24

16. Primary Outcome: Number of Participants Having Normal Fasting Baseline Glucose Value With Treatment-Emergent High Fasting Glucose at Any Time Post Baseline
Description: Normal to high fasting glucose ≤100 milligrams per deciliter (mg/dL) at baseline to ≥126 mg/dL any time post baseline.
Time Frame: Randomization to end of study up to 76 months
Population: Participants with normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 864
participants | 20

17. Primary Outcome: Number of Participants Having Normal Fasting Baseline Lipid Value With Treatment-Emergent High Fasting Lipid at Any Time Post Baseline
Description: Normal to high fasting total cholesterol ≤200 mg/dL at baseline to ≥240 mg/dL any time post baseline. Fasting triglycerides <150 mg/dL at baseline to ≥200 mg/dL and <500 mg/dL any time post baseline.
Time Frame: Randomization to end of study up to 76 months
Population: Participants with normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
participants
  Cholesterol (n=873) | 28
  Triglycerides (n=879) | 41

18. Primary Outcome: Change From Baseline in Weight at Month 76 Endpoint
Description: Mean change in weight from baseline to last observation carried forward (LOCF) endpoint.
Time Frame: Baseline, up to 76 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 919
kilogram (kg) | 2.10 (7.81)

19. Primary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Weight Gain at Month 76 Endpoint
Description: PCS weight gain is defined as a ≥7% increase in weight from baseline.
Time Frame: Randomization to end of study up to 76 months
Population: Participants with normal baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 919
participants | 373

20. Primary Outcome: Number of Participants With Extrapyramidal Symptoms at Any Time
Description: Extrapyramidal symptoms are defined as Simpson-Angus total score (SAS) >3 at any post-baseline visit; Barnes Akathisia Scale (BAS) global score ≥2 at any post-baseline visit; A score ≥3 for any of Abnormal Involuntary Movement Scale (AIMS) for items 1-7 or a score ≥2 for any two of these items. Score for SAS is 0-4 for each of the 10 questions, with 0=normal and 4=extreme. The possible total score for SAS is 0-40. Possible score for BAS is 0-5, with 0=absent and 5=sever. Score 0-4 for each item of AIMS, with 0 =none and 4= sever. Possible total score for items 1-7 is 0-28.
Time Frame: Randomization to end of study up to 76 months
Population: Participants with a baseline and at least one post-baseline measurement.
Measure: Number; unit: participants
Arm/Group | Intramuscular Olanzapine Depot
Number analyzed (Participants) | 931
participants
  SAS (n=819) | 66
  BAS (n=856) | 34
  AIMS (n=860) | 28

ADVERSE EVENTS:
Arm/Group | Intramuscular Olanzapine Depot
Serious Adverse Events (participants affected / at risk) | 170/931
Other Adverse Events (participants affected / at risk) | 501/931
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramuscular Olanzapine Depot (N=931)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiomyopathy alcoholic (Cardiac disorders) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Malaise (General disorders) | 3 (3)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Breast cellulitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3)
Ear infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Leptospirosis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 3 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (4)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 1 (2)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (2)
Coma (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysarthria (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Loss of consciousness (Nervous system disorders) | 2 (2)
Parkinsonism (Nervous system disorders) | 1 (2)
Sedation (Nervous system disorders) | 12 (13)
Somnolence (Nervous system disorders) | 5 (5)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 4 (5)
Agitation (Psychiatric disorders) | 6 (7)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (6)
Completed suicide (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (5)
Delirium (Psychiatric disorders) | 4 (4)
Delusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 5 (5)
Disorientation (Psychiatric disorders) | 1 (2)
Emotional disorder (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 2 (2)
Impulsive behaviour (Psychiatric disorders) | 1 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 5 (5)
Psychotic disorder (Psychiatric disorders) | 20 (21)
Restlessness (Psychiatric disorders) | 1 (2)
Schizophrenia (Psychiatric disorders) | 35 (38)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 8 (9)
Suicide attempt (Psychiatric disorders) | 4 (4)
Vomiting psychogenic (Psychiatric disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3)
Social stay hospitalisation (Social circumstances) | 1 (1)
Plastic surgery (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramuscular Olanzapine Depot (N=931)
Nasopharyngitis (Infections and infestations) | 74 (84)
Weight increased (Investigations) | 134 (136)
Dizziness (Nervous system disorders) | 50 (57)
Headache (Nervous system disorders) | 67 (72)
Somnolence (Nervous system disorders) | 85 (101)
Anxiety (Psychiatric disorders) | 90 (94)
Depression (Psychiatric disorders) | 48 (48)
Insomnia (Psychiatric disorders) | 90 (92)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days